CLINICAL TRIAL: NCT06024083
Title: Dialectical Behavior Therapy Skills Video Intervention for Chinese and Chinese American College Students
Brief Title: Skills Video Intervention for Chinese/Chinese Americans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Shireen L. Rizvi, PhD, ABPP, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2023001220
Record Dates: First submitted 2023-08-08; First posted 2023-09-05 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Emotion Regulation; Self Efficacy; Acceptability of Health Care
Keywords: Dialectical Behavior Therapy; Ecological Momentary Assessment; Psychotherapy, Brief; Culturally Competent Care
MeSH Terms: conditions — Emotional Regulation; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assessment only (No Intervention): Daily assessment of emotion regulation and self-efficacy variables.
- Acceptance-oriented skills followed by change-oriented skills (Experimental): Administration of acceptance-oriented skills videos first followed by change-oriented skills videos.
  Interventions: Behavioral: Dialectical Behavior Therapy skills video intervention
- Change-oriented skills followed by acceptance-oriented skills (Experimental): Administration of change-oriented skills videos first followed by acceptance-oriented skills videos.
  Interventions: Behavioral: Dialectical Behavior Therapy skills video intervention

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy skills video intervention — A series of 14 animated videos (9 acceptance-oriented and 5 change-oriented skills videos) available in both English and Mandarin Chinese.
  Arms: Acceptance-oriented skills followed by change-oriented skills; Change-oriented skills followed by acceptance-oriented skills

SUMMARY:
This is a study that aims to test a coping skills intervention delivered via brief animated videos for Chinese and Chinese American college students.

DETAILED DESCRIPTION:
We are interested in seeing whether a brief video-based Dialectical Behavior Therapy skills training intervention that incorporates Western psychotherapy components and Eastern philosophies would be perceived as relevant and useful for this culturally unique yet diverse group. During the study, participants will (1) complete a 20-min online baseline questionnaire; (2) complete a brief survey each day using a phone App for up to four weeks; and may (3) receive a video each day during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* identifying as Chinese or Chinese American
* interested in learning coping skills to regulate emotions
* having a smart-phone compatible with the research mobile phone app
* matriculated at the local University for the current semester

Exclusion Criteria:

* currently receiving routine mental health services
* not able to read or write English
* not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Emotion regulation measured by a combination of questions | daily for up to 4 weeks
  A combination of questions on emotional states, context for emotions, how intolerable and distressing emotions are, use of emotion regulation strategies, perceived effectiveness of emotion regulation, and Patient-Reported Outcomes Measurement Information System Self-efficacy of Managing Emotions Short-form 4a (a 4-item measure of the confidence to manage emotional states rated using a 5-point Likert scale)
General self efficacy measured by Patient-Reported Outcomes Measurement Information System General Self-Efficacy Short-form 4a | daily for up to 4 weeks
  A 4-item measure of the ability to successfully perform specific tasks and behaviors rated using a 5-point Likert scale
Acceptability/usability of intervention measured by a combination of Likert-scale and open-ended questions | daily following the delivery of each video for up to 2 weeks
  A combination of questions that involve rating the acceptability and usability of skills videos (e.g., "how useful do you think the skills will be") and open-ended questions on cultural relevance

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Yin, M.S., Study Director — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT06024083/ICF_000.pdf